CLINICAL TRIAL: NCT04968171
Title: Assessment of Physical Effort in People With Newly Diagnosed Type 1 Diabetes Mellitus and Its Impact on: Partial Clinical Remission, Insulin Resistance, HDL Cholesterol Function, Immune Function and Length of Life.
Brief Title: Diabetes Type 1 and Fitness.
Acronym: Diab1Fit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 1050/19
Record Dates: First submitted 2020-08-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus type 1; Physical activity; Clinical remission
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with newly diagnosed diabetes mellitus type 1: People with newly diagnosed diabetes mellitus type 1 admitted to the Department of Internal Medicine and Diabetology.
  Treated with intensive insulin therapy. Measurement of VO2max between 3 and 12 month after diagnosis. Further continuous observation with follow-up every year and evaluation of final end-points after 5 and 10 years.

SUMMARY:
The Diab1Fit Study project aims to a multidirectional assessment of physical activity and its impact in people with type 1 diabetes (DM1). To the study are recruited people with newly diagnosed DM1, treated with intensive functional insulin therapy from the beginning of the disease. The study is planned to cover a minimum of 100 people with newly diagnosed DM1 and lead prospective observation of this group (for a minimum of 5-10 years). The investigators will evaluate the effect of VO2max in people with newly diagnosed DM1 on partial clinical remission. What is more the investigators also assess quantitative and qualitative changes of plasma lipoproteins, with particular emphasis on HDL metabolism, mechanism linking VO2max with management of DM1 (longevity proteins, miostatin, insulin resistance) and immune function.

DETAILED DESCRIPTION:
The Diab1Fit Study project aims to a multidirectional assessment of physical activity and its impact in people with type 1 diabetes (DM1). To the study are recruited people with newly diagnosed DM1, treated with intensive functional insulin therapy from the beginning of the disease. The study is planned to cover a minimum of 100 people with newly diagnosed DM1 and lead prospective observation of this group (for a minimum of 5-10 years). The investigators will evaluate the effect of VO2max in people with newly diagnosed DM1 on partial clinical remission. What is more the investigators also assess quantitative and qualitative changes of plasma lipoproteins, with particular emphasis on HDL metabolism, mechanism linking VO2max with management of DM1 (longevity proteins, miostatin, insulin resistance) and immune function.

Patients will be assessed: during the first hospitalization in the moment of diagnosis (prior to introduction of insulin treatment), after 3 weeks, after 6 months and after 12 months of insulin therapy. Further observations planned in the annual intervals. Further continuous observation with follow-up every year and evaluation of final end-points after 5 and 10 years. In addition, the study group will be under constant monitoring of metabolic evaluation every three months in the Outpatient Clinic. An additional visit to assess VO2max will be scheduled between 3 and 12 months of diabetes. The investigators will use an ergospirometer (COSMED K5 System) during an exercise test carried out on a cycloergometer (progressive exercise test). Moreover, the investigators will monitor glucose levels during the exercise test - using a continuous glucose monitoring system using the FreeStyle Libre Flash Glucose Monitoring System (Abbott). A week before the exercise test, the investigators will borrow a Garmin watch that assesses the patient's daily activities

During each follow-up will be assessed parameters:

1. The presence of partial clinical remission, according to Mortensen: HbA1c (%) + [4 x dawka insuliny (j/kg/d)] ≤ 9.
2. Data on lifestyle (diet, exercise), family history and smoking.
3. Anthropometric data:

   1. BMI (body mass index) = weight [kg]/(height [m])2
   2. Waist circumference
   3. WHR - waist to hip ratio
   4. daily insulin requirement (U/kg m.c./d),
   5. eGDR (estimated glucose disposal rate) = 24.31-12.22(WHR)-3.29(hypertension 0/1)-0.57( HbA1c [mg/kg/min])
   6. VAI (visceral adiposity index):

      For women = [Waist circumference/36.58+(1.89xBMI)]x(TG/0.81)x(1.52/HDL), For men = [Waist circumference /39.68+(1.88xBMI)]x(TG/1.03)x(1.31/HDL),
   7. body composition analysis
4. Parameters of diabetes metabolic control

   1. Lipid profile
   2. Glycated hemoglobin level (HbA1c)
5. Protein glycation end products Expected impact of the research project on the development of science, civilization and society: The study confirms the great importance of aerobic physical activity in the treatment of people with DM1 from the beginning of the diagnosis. The project aims to pay attention to the importance of physical activity among people with DM1 and to popularize this method of treatment. The obtained results will be used for the prospective observation of this group to assess the impact of physical effort on the development of chronic complications and will allow planning intervention studies in this population. The results of this study will help enrich knowledge about the body's ability to exercise among people with DM1 and show new intervention solutions. It may contribute to changing the recommendations of scientific societies. What is more knowledge about prolonging partial clinical remission and thereby reducing the risk of developing chronic complications will contribute to the introduction of new recommendations. Research on exercise in diabetes and longevity proteins will increase the length and quality of life of people with DM1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years,
* New onset type 1 diabetes (confirmed by the presence of antibodies - antyGAD, ICA, IA2)
* Treatment with intensive insulin therapy,
* Written consent to participate in the study.

Exclusion Criteria:

* Contraindications to the exercise test (including: recent myocardial infarction, unstable coronary artery disease, hypertrophic cardiomyopathy, serious arrhythmias, myocarditis, advanced systemic diseases, hyperthyroidism, recurrent anemia),
* Mental disorders,
* Co-morbidities with potential impact on physical performance (e.g. cancer, renal failure, liver failure, rheumatic diseases, COPD, asthma, anemia, hypothyroidism and hyperthyroidism),
* Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A minimum of 100 people with newly diagnosed type 1 diabetes hospitalized in the Department of Internal Medicine and Diabetology Poznan University of Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VO2max [ml/min/kg] | 1 year
  VO2 max level evaluated during ergospirometry (COSMED K5)
Partial clinical remission time | 1 year
  Presence [(4 x insulin dose (j/kg/d)] ≤ 9] and duration [time] of partial clinical remission

SECONDARY OUTCOMES:
Triglicerydes concentriation in serum [mg/dl] | Change from baseline in apolipoproteins' at 6 and 12 months
  Changes in serum triglyceride levels
LDL-C concentriation in serum [mg/dl] | Change from baseline in apolipoproteins' at 6 and 12 months
  Changes in serum LDL levels
HDL-C concentriation in serum [mg/dl] | Change from baseline in apolipoproteins' at 6 and 12 months
  Changes in serum HDL levels
Total Cholesterol concentriation in serum [mg/dl] | Change from baseline in apolipoproteins' at 6 and 12 months
  Changes in serum Total-CH levels
Lipid tissue content [%] | 5 years
  Evaluation of lipid tissue content prior to yearly visit.
A1c [%] | 5 years
  Changes in serum A1c levels
Daily insulin requirement [u/kg/d] | 1 year
  Sum of insulin units administered in the day prior to yearly visit.
Retinopathy | 5 years
  Evaluation of retinopathy (ophthalmology assessment)
Neuropathy | 5 years
  Evaluation of presence of neuropathy peripheral and autonomic (clinical examination, Visual Analog Score for pain and ProsciCard)
eGFR [ml/min/1,73m2] | 5 years
  Assessment of glomerular filtration and renal filtration function
Creatynine [mg/dl] | 5 years
  Assessment of renal function
Albumine to creatynine ratio ACR [mg/g] | 5 years
  Assessment of renal function

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine and Diabetiology Poznan University of Medical Sciences, Poznan, Poland